CLINICAL TRIAL: NCT06637930
Title: Clinical and Radiographic Evaluations of Implant Retained Mandibular Overdenture Using CAD\CAM Fabricated Telescopic Crown: Randomized Clinical Trial
Brief Title: Comparing Cobalt-Chromium Versus PEEK Secondary Telescopic Crowns on Implant Retained Mandibular Overdenture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amr El Sayed Khalifa (Other)
Responsible Party: Sponsor-Investigator, Amr El Sayed Khalifa, assistant lecturer of prosthodontics, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 528
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Edentulism

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cobalt chromium(COCR) group (Experimental): The secondary crowns and the framework were fabricated using milled Cobalt chromium alloy
  Interventions: Other: Edentulous Alveolar Ridge In Mandible
- Polyetheretherketone(PEEK) Group (Experimental): The secondary crowns and the framework were fabricated using milled PEEK material
  Interventions: Other: Edentulous Alveolar Ridge In Mandible

INTERVENTIONS:
Other: Edentulous Alveolar Ridge In Mandible — implant retained mandibular overdenture using telescopic attachment system. all the patients received 2 implants at the canine region bilaterally using sterelithographic guide , then healing period for 3 months for proper osseointegration , then digital intraoral scanning was performed to detect implant position using scannable bodies , abutments which act as primary crowns were designed on cad software then milled using premilled titanium abutments.the study grouping was performed then virtual model was done for the designing of the frameworks then milled according to the grouping of the study. Try in of the frameworks was done and overdentures were inserted.
  * Retention force test was done using digital force gauge.
  * Probing depth using Teflon coated periodontal probe.
  * Marginal bone level and bone density were measured using digital periapical x-ray

SUMMARY:
The aim of this randomized clinical trial was to compare

I- The clinical behavior of implant retained removable overdenture using telescopic retention system fabricated using CAD\CAM techniques where the effects of the different material combinations were examined in regard to:

1. Retention of the mandibular over-denture.
2. Plaque accumulation, presence of calculus, bleeding tendency, health of peri-implant mucosa and probing depth.

II - The radiographic behavior regarding marginal bone level and bone density.

DETAILED DESCRIPTION:
This study compared implant-retained telescopic mandibular overdentures reinforced with milled metal framework (Co-Cr) and milled polymer (PEEK) in terms of retention, periimplant mucosal health, and radiographic changes in twelve patients.

Initially, all patients received conventional complete dentures. A CBCT was conducted prior to the implant surgical phase using a radiographic stent. Two implants were inserted interforaminally using a flapless method. The implants were then left for three months to allow for osseointegration, and the patients were instructed to wear their complete dentures during the healing process.

Following the osseointegration period, the prosthetic phase began, with all patients obtaining primary crowns constructed from titanium alloys. The patients were then randomly divided into two groups, 6 patients in each group. Group A received a COCR framework that included secondary crowns while group B received a PEEK framework and secondary crowns.

Retention was tested for each group (baseline, 6 months, 9 months, and 12 months) using a digital force gauge. The pulling force gradually increased until the denture was dislodged. The retentive force was measured during the initial separation of the telescopic crown.

Soft tissue conditions was assessed using single coded probe for each group (baseline, 6 months, 9 months, and 12 months).Bleeding tendency on probing, plaque accumulation, calculus deposition, perimplant mucosal health were the parameters for each group evaluation.

While the radiographic assessment was performed for each group (baseline, 6months, 9 months and12 months) using digital periapical radiographs by the means of XCP instrument and digital sensor. The marginal bone level was measured by evaluating the difference of bone level at the neck of the implant. The bone density was evaluated at three areas surrounding the implants.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients
* Absence of any systematic contraindications to implant surgery,
* Presence of sufficient bone height and width to accommodate implants with length 14mmm and diameter 3.6mm.
* Inter-arch distance more than or equal 10 mm.
* Four months since the last extraction had taken place.
* No previous bone augmentation procedures.

Exclusion Criteria:

* psychological disorders prohibiting implant treatment.
* Heavy smoking (10 cigarettes/day)
* Alcohol and/or drug abuse,
* Physical disability that may interfere with the ability to perform oral hygiene.
* Patients were receiving drugs which impair healing .

Ages: 52 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
intraoral retention force assessment in Newtons (N) | 1 year follow up
  using force gauge at the geometric center of the overdentiure

OTHER OUTCOMES:
Probing depth in millimeters(mm) | 1 year follow up
  using periodontal probe
Radioghraphic marginal bone level measurement in millimeters (mm) | 1 year
  using digital peri-apical x rays in a paralleling technique using XCP device

CONTACTS AND LOCATIONS:
Overall Officials: Emad TB Agamy, Professor of Prosthodontics, Study Chair — Faculty of Dentistry, Minia university
Locations (1):
- Faculty of Dentistry, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No